CLINICAL TRIAL: NCT01529775
Title: A Prospective Randomized-controlled Evaluation of the Osseotite Certain Tapered Prevail Implant for the Preservation of Crestal Bone
Brief Title: Randomized Study of Osseotite Certain Tapered Prevails vs. Osseotite Certain Tapered
Acronym: Bolivar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ZimVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3008
Record Dates: First submitted 2012-02-07; First posted 2012-02-09 (Estimated); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Partial Edentulism; Tooth Disease
Keywords: partial edentulism; dental implants; Osseotite Certain Prevail Tapered; Osseotite Certain Tapered; Crestal bone level; randomized; clinical study
MeSH Terms: conditions — Tooth Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Osseotite Certain Tapered Prevail (Experimental): Osseotite Certain Tapered Prevail design with platform switching feature
  Interventions: Device: Osseotite Certain Tapered Prevail
- Osseotite Certain Tapered (Active Comparator): Osseotite Certain Tapered implant with non-platform switching design
  Interventions: Device: Osseotite Certain Tapered

INTERVENTIONS:
Device: Osseotite Certain Tapered Prevail — Osseotite implant with platform switching feature
  Other Names: Osseotite endosseous dental implant
  Arms: Osseotite Certain Tapered Prevail
Device: Osseotite Certain Tapered — Osseotite implant with non-platform switching feature
  Other Names: Osseotite endosseous dental implant
  Arms: Osseotite Certain Tapered

SUMMARY:
This study will demonstrate the benefits of platform switching design of the Osseotite dental implant.

DETAILED DESCRIPTION:
The Osseotite Certain Prevail implant with its platform switch feature will demonstrate higher success rate than the non-platform Osseotite Certain implant

ELIGIBILITY:
Inclusion Criteria:

* patients of either sex and older than 18 years of age
* patients needing at least one dental implant to treat partial edentulism
* patients physically able to tolerate surgical and restorative dental procedures
* patients agreeing to all protocol visits

Exclusion Criteria:

* patients with infection or severe inflammation at the intended treatment sites
* patients smoking greater than 10 cigarettes per day
* patients with uncontrolled diabetes mellitus
* patients with uncontrolled metabolic diseases
* patients who received radiation treatment to the head in the past 12 months
* patients needing bone grafting at the intended treatment sites
* patients known to be pregnant at screening visit
* patients with para-functional habits like bruxing and clenching

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2010-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Cumulative Success Rate | 3 years
  An implant will be considered successful if it is immobile when tested at various study time point

SECONDARY OUTCOMES:
Crestal Bone Regression | 3 years
  Differences in crestal bone levels obtained at various study time points will be compared between the two implant designs

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Pavez, DDS, Principal Investigator — Universidad Finis Terrae
Locations (1):
- Universidad Finis Terrae, Santiago, Chile

IPD SHARING:
Plan to Share IPD: No